CLINICAL TRIAL: NCT05992428
Title: An Open-label, 2-Part, Phase 1 Clinical Trial to Evaluate Drug Interactions When DA-8010 is Co-administered With Paroxetine or Mirabegron in Healthy Adults
Brief Title: Drug Interactions When DA-8010 is Co-administered With Paroxetine or Mirabegron in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA8010_DIPM_I
Record Dates: First submitted 2023-07-27; First posted 2023-08-15 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — DA-8010; Paroxetine; mirabegron

STUDY DESIGN:
Intervention Model Description: 2-part
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1 or 2 (Experimental): [Part 1] DA-8010 5mg + Paroxetine 20mg [Part 2] DA-8010 5mg + Mirabegron 50mg
  Interventions: Drug: DA-8010 5mg; Drug: Paroxetine 20mg; Drug: Mirabegron 50mg

INTERVENTIONS:
Drug: DA-8010 5mg — [Part 1] DA-8010 5mg + Paroxetine 20mg [Part 2] DA-8010 5mg + Mirabegron 50mg
Drug: Paroxetine 20mg — [Part 1] DA-8010 5mg + Paroxetine 20mg
Drug: Mirabegron 50mg — [Part 2] DA-8010 5mg + Mirabegron 50mg

SUMMARY:
This is an open-label, 2-Part, phase 1 study to evaluate drug interactions when DA-8010 is co-administered with Paroxetine or Mirabegron in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteer 19 years to 50 years
* Body weight in the range of 40.0 to 90.0 kg and body mass index in the range of 18 to 28kg/m2
* The subjects personally signed and dated informed consent document after informed of all patient aspects of the study, fully understanding and determined spontaneously to participate
* In the case of female volunteers, those who are not necessarily pregnant or lactating or who are in a surgical infertility condition (both tubular obstruction, hysterectomy, bilateral tubular resection, etc.)
* The subjects who are judged appropriate to participate this clinical trial according to the physical examination, routine laboratory examination and questionnaire

Exclusion Criteria:

* Subject with serious active hepatobiliary (severe hepatic failure, etc.), renal(severe renal impairment, etc.), neurologic, immunologic, respiratory, digestive, endocrine, hematologic, cardiovascular(heart failure, Torsades de pointes, etc), urologic, psychological disease or history of such disease
* Subject with gastrointestinal disease (peptic ulcer, gastritis, gastrospasm, gastroesophageal reflux disease, Crohn's disease, etc.) or history of such disease/surgery (excluding simple appendic surgery, hernia surgery, hemorrhoid surgery)
* Subject Hypersensitive to any of the IP components or other drug components(Aspirin, Antibiotics, etc.)
* Subject who is positive for serum test results (hepatitis B test, hepatitis C test, HIV test, syphilis test)
* Subject who have history of drug/alcohol abuse or Positive in Urine drug screen test
* Subject who determined that Investigator is unfit to participate in a clinical trial due to other reasons other than the above items

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 0~48hours
  PK Parameter
Area under the plasma concentration versus time curve of DA-8010 (AUClast) | 0~48hours
  PK Parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Soeul, South Korea